CLINICAL TRIAL: NCT01107444
Title: A Randomized Phase 2 Study of LY2181308 in Combination With Docetaxel Versus Docetaxel in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Were Previously Treated With First Line Chemotherapy
Brief Title: Study of LY2181308 in Combination With Docetaxel Versus Docetaxel in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11766; H8Z-MC-JACW (Other: Eli Lilly and Company); 2009-017591-24 (EudraCT Number)
Record Dates: First submitted 2010-04-15; First posted 2010-04-21 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; LY 2181308

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2181308 + Docetaxel (Experimental): LY2181308: 750 milligrams (mg), intravenous (IV), on Day -2 and Day -1 of a 2 day lead-in period; on Day 1, Day 6, and Day 14 for Cycle 1 (1 cycle = 21 days); and once weekly for Days 1 through 21 for Cycles 2 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met.
  Docetaxel: 75 milligrams/square meter (mg/m^2), intravenous (IV), on Day 1 of Cycle 1 (1 cycle = 21 days) and on Day 1 of Cycles 2 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met.
  Interventions: Drug: Docetaxel; Drug: LY2181308
- Docetaxel (Active Comparator): Docetaxel: 75 milligrams/square meter (mg/m^2), intravenous (IV) on Day 1 of Cycles 1 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Administered intravenously
Drug: LY2181308 — Administered intravenously
  Arms: LY2181308 + Docetaxel

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of LY2181308 in combination with docetaxel compared to docetaxel alone in participants with non-small cell lung cancer who were previously treated with first line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-small cell lung cancer with locally or advanced metastatic disease(Stage IIIB or IV at entry) not amenable to curative therapy and who have progressed after 1 line of chemotherapy
* Measureable disease as defined by response evaluation criteria in solid tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Must make available any existing tumor tissue from the primary biopsy
* Participants with prior radiation may be eligible if they meet certain criteria
* Adequate bone marrow reserve and organ functioning
* Women must have a negative pregnancy test and must comply with a highly reliable contraceptive method during and for 6 months after the treatment period and must not be breastfeeding
* Men must comply with a contraceptive regimen during and for 6 months after the treatment period

Exclusion Criteria:

* Currently enrolled in or discontinued a clinical trial involving an investigational drug/device within the last 30 days. Participants may be permitted to enter treatment before the 30 day waiting period in special circumstances
* Pregnant or breastfeeding
* Serious concomitant systemic disorders that would compromise the safety of the participant or the participant's ability to complete the study
* Second primary malignancy that could affect compliance with the protocol or interpretation of the study results
* Known allergy or hypersensitivity to docetaxel, taxanes, LY2181308, oligonucleotides, or any component of the formulations
* Participants with documented central nervous system or brain metastasis at the time of study entry
* Pre-existing neuropathy equivalent to a common terminology criteria for adverse events(CTCAE)code greater than or equal to 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lebanon, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braunschweig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karlsruhe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aviano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lido di Camaiore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin-Zdunowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, England
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Headington, Oxford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, Trent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Natale R, Blackhall F, Kowalski D, Ramlau R, Bepler G, Grossi F, Lerchenmuller C, Pinder-Schenck M, Mezger J, Danson S, Gadgeel SM, Summers Y, Callies S, Andre V, Das M, Lahn M, Talbot D. Evaluation of antitumor activity using change in tumor size of the survivin antisense oligonucleotide LY2181308 in combination with docetaxel for second-line treatment of patients with non-small-cell lung cancer: a randomized open-label phase II study. J Thorac Oncol. 2014 Nov;9(11):1704-8. doi: 10.1097/JTO.0000000000000285. PMID 25436803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Started | 120 | 60
Received At Least 1 Dose of Study Drug | 114 | 48
Completed | 112 | 47
Not Completed | 8 | 13
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Protocol Entry Criteria Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2181308 + Docetaxel | Docetaxel | Total
Number analyzed (Participants) | 114 | 48 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.19 (9.74) | 64.10 (8.37) | 62.05 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 16 | 59
  Male | 71 | 32 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 110 | 45 | 155
  Black or African American | 3 | 3 | 6
  Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 12 | 45
  Poland | 20 | 9 | 29
  Belgium | 5 | 0 | 5
  Germany | 17 | 10 | 27
  Italy | 15 | 3 | 18
  United Kingdom | 24 | 14 | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) classifies participants according to their functional impairment. Scores range from 0 (Fully Active), 1 (Ambulatory, restricted strenuous activity) to 5 (Death). For inclusion in this study, participants had an ECOG PS of 0 to 1.
  Participants
    0 | 37 | 13 | 50
    1 | 77 | 35 | 112
Initial pathological diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma, poorly differentiated, lung | 1 | 0 | 1
  Adenocarcinoma, bronchioalveolar | 5 | 0 | 5
  Adenocarcinoma, lung | 58 | 20 | 78
  Neuroendocrine carcinoma (CA) | 1 | 0 | 1
  Large cell lung CA | 1 | 0 | 1
  Non-small cell lung carcinoma (NSCLC) | 14 | 4 | 18
  NSCLC, poorly differentiated | 9 | 0 | 9
  Squamous cell lung CA | 25 | 23 | 48
  NSCLC, not otherwise specified (NOS) | 0 | 1 | 1
Disease stage at study entry [Count of Participants; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes; Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver
  Participants
    Stage IIIB | 10 | 6 | 16
    Stage IV | 104 | 42 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tumor Size to the End of Cycle 2
Description: The tumor size was defined as the sum of the longest diameters for the target lesions. The sum of lesion diameters was calculated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. The log ratio of tumor size at the end of Cycle 2 to tumor size at baseline was calculated for each participant.
Time Frame: Baseline, End of Cycle 2 (1 cycle = 21 days)
Population: Participants who received at least 1 dose of study drug and had tumor size measurements (according to the pre-specified inclusion criteria) at baseline and at the end of Cycle 2.
Measure: Mean (Standard Deviation); unit: Log Ratio of Tumor Size
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 82 | 42
Log Ratio of Tumor Size | 1.06 (0.2) | 1.01 (0.13)
Statistical Analysis 1: Comparison: LY2181308 + Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.284, t-test, 1 sided — The t-test was based on the logarithm of the ratio of tumor size at Cycle 2 to that at baseline as this measure follows a normal distribution

2. Secondary Outcome: Number of Participants With Characterization of Toxicities as Defined by Common Terminology Criteria for Adverse Events (CTCAE) Coding
Description: Safety analyses included listings and/or summaries of the following:
  1. CTCAE for laboratory and non-laboratory parameters possibly related to study drug;
  2. CTCAE Grades 3 and 4 for laboratory and non-laboratory parameters possibly related to study drug (Grade 3 - severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care. Grade 4 - life-threatening consequences; urgent intervention indicated);
  3. Dose adjustments due to adverse events (AEs).
Time Frame: Randomization through long-term follow up (up to 21.6 months)
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Participants
  Participants with >= 1 CTCAE | 98 | 42
  Participants with >= 1 CTCAE Grade 3 or Grade 4 | 76 | 34
  Participants with Docetaxel Dose Changes Due to AE | 24 | 11
  Participants with LY2181308 Dose Changes Due to AE | 8 | NA — Participants in this arm of the study did not receive LY2181308.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from date of first dose to the first observation of disease progression or death due to any cause. PFS time was censored at the date of the last assessment visit for participants who were still alive and who did not have documented progressive disease as of the data cut-off date.
Time Frame: Randomization to the first date of progressive disease or death from any cause (up to 12.88 months)
Population: Participants who received at least 1 dose of study drug. A total of 10 participants were censored in the Docetaxel arm; 18 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Months | 2.83 [1.84 to 3.65] | 3.35 [2.69 to 4.57]

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve From Zero to 4 Hours (AUC[0-4]) for LY2181309 and Docetaxel
Description: Pharmacokinetics: Area Under the Concentration Curve From Zero to 4 hours (AUC[0-4]) for LY2181309 and Docetaxel
Time Frame: Docetaxel: Cycle(C)1 Day(D)1:0,1,1.25,1.75,3,4 hours(h);LY2181308 + Docetaxel: C1 D-1:3,4 h;D1:0,3,4 h
Population: Participants who received at least 1 dose of study drug and who had an interpretable pharmacokinetic profile
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- LY2181308 + Docetaxel: LY2181308: 750 milligrams (mg), intravenous (IV), on Day -2 and Day -1 of a 2 day lead-in period; on Day 1, Day 6, and Day 14 for Cycle 1 (1 cycle = 21 days); and once weekly for Days 1 through 21 for Cycles 2 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met.
  Docetaxel: 75 milligrams/meters squared (mg/m^2), intravenous (IV), on Day 1 of Cycle 1 (1 cycle = 21 days) and on Day 1 of Cycles 2 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met.
- Docetaxel: Docetaxel: 75 milligrams/meters squared (mg/m^2), intravenous (IV) on Day 1 of Cycles 1 through 6 (1 cycle = 21 days). After 6 cycles, it was possible to continue therapy until progression of disease, unacceptable toxicity, or another withdrawal criterion was met
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 85 | 42
nanograms*hours per milliliter (ng*h/mL) | 1642 (76.4) | 1195 (104)

5. Secondary Outcome: Pharmacokinetics: Area Under the Drug Concentration-Time Curve From Zero to Infinity (AUC[0 ∞]) of LY2181309 and Docetaxel
Description: Pharmacokinetics: Area Under the Drug Concentration-Time Curve From Zero to Infinity (AUC[0 ∞]) of LY2181309 and Docetaxel
Time Frame: Docetaxel: Cycle(C)1 Day(D)1:0,1,1.25,1.75,3,4,5,505,513,2521 hours(h);LY2181308 + Docetaxel: C1 D -1:3,4 h;D1:0,3,4,5,5.25,5.75,7,8,120,504,507,509,1008,1512,1515,1517,2016, 2520,2523,2525 h
Population: Participants who received at least 1 dose of study drug and who had an interpretable pharmacokinetic profile
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 85 | 42
nanograms*hours per milliliter (ng*h/mL) | 1905 (64.7) | 1778 (87.8)

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was the duration from enrollment to death from any cause. For participants who were alive, OS is censored at the date of last contact.
Time Frame: Randomization to date of death from any cause (up to 21.6 months)
Population: Participants who received at least 1 dose of study drug. A total of 20 participants were censored in the Docetaxel arm; 41 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
months | 7.9 [6.6 to 9.7] | 8.8 [5.7 to 13.8]

7. Secondary Outcome: Time to Worsening of Symptoms as Defined by Lung Cancer Symptom Score (LCSS) Questionnaire
Description: The worsening of symptoms was defined as a 15-millimeter (mm) increase in any 1 symptom on the LCSS. The LCSS is an assessment used to evaluate 6 major symptoms associated with lung malignancies and their effect on overall symptomatic distress, functional activities, and global quality of life. LCSS consists of 2 scales: 1 completed by the participant and 1 completed by the health care professional (which is the average symptom burden index [ASBI]). Participant-reported outcomes are assessed using 9 visual analog scales (100-mm horizontal line). Participants indicate intensity of response to the items in question (0 = lowest rating, 100 = highest rating). The LCSS total score ranges from 0 (lowest rating) to 100 (highest rating). The LCSS total score was defined as the mean over all 9 items. Time to worsening of symptoms was censored at the date of the last assessment visit for participants who did not experience any worsening of symptoms as of the data cut-off date.
Time Frame: Baseline to the worsening of symptoms (up to 4.6 months)
Population: Participants who received at least 1 dose of study drug. A total of 10 participants were censored in the Docetaxel arm; 26 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Months | 1.0 [0.7 to 1.0] | 0.8 [0.5 to 1.1]

8. Secondary Outcome: Time to Objective Tumor Response of Partial Response (PR) or Complete Response (CR)
Description: Time to objective tumor response was defined as the time from the date of randomization to the first date of documented objective tumor response. Time to objective tumor response was censored at the date of the last assessment visit for participants who had not had documented response as of the data cut-off date. Complete response (CR) was defined as the disappearance of all target lesions; partial response (PR) was defined as at least a 30% decrease in sum of the longest diameter of target lesions.
Time Frame: Randomization to the date of first response (up to 12.1 months)
Population: Participants who received at least 1 dose of study drug. A total of 47 participants were censored in the Docetaxel arm; 107 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Months | NA [NA to NA] — Due to the high rate of censored participants (107 of 114 participants), the median could not be calculated. | NA [NA to NA] — Due to the high rate of censored participants (47 of 48 participants), the median could not be calculated.

9. Secondary Outcome: Time to Documented Disease Progression
Description: Time to documented disease progression was defined as the time from the date of randomization to the first date of documented progression. Progressive disease (PD) was defined as at least a 20% increase in sum of longest diameter of target lesions. Time to documented disease progression was censored at the date of the last assessment visit for participants who had not had documented progressive disease as of the data cut-off date.
Time Frame: Randomization to the first date of progressive disease (up to 12.9 months)
Population: Participants who received at least 1 dose of study drug. A total of 15 participants were censored in the Docetaxel arm; 38 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Months | 2.9 [2.0 to 3.7] | 3.4 [2.8 to 5.6]

10. Secondary Outcome: Percent of Participants Having a Partial Response (PR) or a Complete Response (CR)
Description: Complete response (CR) was defined as the disappearance of all target lesions; partial response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Randomization to the first date of progressive disease (up to 12.1 months)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 114 | 48
Percentage of participants | 6.1 | 2.1

11. Secondary Outcome: Duration of Response
Description: Duration of response was measured from the time measurement criteria were met for complete response (CR) or partial response (PR) (whichever was first recorded) until the first date of documented progressive disease (PD) or death. Complete response (CR) was defined as the disappearance of all target lesions; PR was defined as at least a 30% decrease in sum of longest diameter of target lesions; PD was defined as at least a 20% increase in sum of longest diameter of target lesions. Duration of response was censored at the date of the last assessment or follow-up visit for responders who were still alive and had not progressed.
Time Frame: Time of response to progressive disease (PD) (approximately 8.7 months)
Population: Participants who received at least 1 dose of study drug and achieved CR or PR. A total of 0 participants were censored in the Docetaxel arm; 2 participants were censored in the LY2181308 + Docetaxel arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 5 | 1
Months | 2.8 [2.8 to NA] — The upper range of the confidence interval (CI) could not be calculated due to lack of data (5 response events, 2 participants censored). | 5.4 [NA to NA] — The confidence interval (CI) could not be calculated due to lack of data (1 response event, 0 participants censored).

12. Secondary Outcome: Lung Cancer Symptom Scale (LCSS) Average Symptom Burden Index (ASBI) on Cycle 2 Day 1
Description: The worsening of symptoms was defined as a 15-millimeter (mm) increase in any 1 symptom on the Lung Cancer Symptom Scale (LCSS). The LCSS is an assessment used to evaluate 6 major symptoms associated with lung malignancies and their effect on 3 overall symptomatic items: distress, functional activities and global quality of life. LCSS consists of 2 scales: 1 completed by the participant and 1 completed by the health care professional (which is the average symptom burden index [ASBI]). Participant-reported outcomes are assessed using 9 visual analog scales (100-mm horizontal line). Participants indicate intensity of response to the items in question (0 = lowest rating, 100 = highest rating). The LCSS total score ranges from 0 (lowest rating) to 100 (highest rating) and was defined as the mean over all 9 items. ASBI was calculated as the mean of six symptom-specific questions from the LCSS, with scores range from 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Cycle 2 Day 1
Population: Participants who received at least 1 dose of study drug and had evaluable LCSS data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 81 | 38
units on a scale | 22 [11 to 34] | 24 [15 to 38]

13. Secondary Outcome: Lung Cancer Symptom Scale (LCSS) Average Total Score at Cycle 2 Day 1
Description: The worsening of symptoms was defined as a 15-millimeter (mm) increase in any 1 symptom on the Lung Cancer Symptom Scale (LCSS). The LCSS is an assessment used to evaluate 6 major symptoms associated with lung malignancies and their effect on 3 overall symptomatic items: distress, functional activities and global quality of life. LCSS consists of 2 scales: 1 completed by the participant and 1 completed by the health care professional (which is the average symptom burden index [ASBI]). Participant-reported outcomes are assessed using 9 visual analog scales (100-mm horizontal line). Participants indicate intensity of response to the items in question (0 = lowest rating, 100 = highest rating). The LCSS total score ranges from 0 (lowest rating) to 100 (highest rating) and was defined as the mean over all 9 items.
Time Frame: Cycle 2 Day 1
Population: Participants who received at least 1 dose of study drug and had evaluable LCSS data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Number analyzed (Participants) | 80 | 37
units on a scale | 27 [11 to 38] | 30 [20 to 41]

ADVERSE EVENTS:
Arm/Group | LY2181308 + Docetaxel | Docetaxel
Serious Adverse Events (participants affected / at risk) | 65/120 | 24/60
Other Adverse Events (participants affected / at risk) | 106/120 | 44/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2181308 + Docetaxel (N=120) | Docetaxel (N=60)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) — Event resulted in death
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal symptom (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Event resulted in death
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 3 (3)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (4) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2181308 + Docetaxel (N=120) | Docetaxel (N=60)
Anaemia (Blood and lymphatic system disorders) | 44 (61) | 13 (16)
Leukopenia (Blood and lymphatic system disorders) | 14 (26) | 10 (27)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 35 (53) | 14 (40)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (20) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (15) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 34 (47) | 22 (28)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 7 (7)
Nausea (Gastrointestinal disorders) | 35 (51) | 12 (14)
Oral pain (Gastrointestinal disorders) | 2 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 13 (13) | 4 (12)
Vomiting (Gastrointestinal disorders) | 23 (31) | 9 (10)
Chest pain (General disorders) | 7 (8) | 3 (3)
Chills (General disorders) | 11 (13) | 0 (0)
Fatigue (General disorders) | 53 (70) | 24 (32)
Mucosal inflammation (General disorders) | 8 (11) | 2 (3)
Oedema peripheral (General disorders) | 13 (16) | 3 (4)
Pain (General disorders) | 1 (1) | 6 (7)
Pyrexia (General disorders) | 26 (33) | 4 (5)
Oral candidiasis (Infections and infestations) | 5 (5) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 24 (33) | 12 (14)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (9) | 4 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (5)
Ageusia (Nervous system disorders) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 6 (6) | 7 (8)
Dysgeusia (Nervous system disorders) | 7 (7) | 7 (7)
Headache (Nervous system disorders) | 10 (11) | 4 (4)
Paraesthesia (Nervous system disorders) | 3 (5) | 3 (5)
Polyneuropathy (Nervous system disorders) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 12 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 33 (33) | 13 (13)
Hypotension (Vascular disorders) | 10 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days